CLINICAL TRIAL: NCT06544954
Title: Assessing Prebiotic Effect of California Grape Consumption on Gut Microbiome and Impact on Intestinal Permeability, Vascular Function, and Systemic Inflammation in Over-weight Subjects: Differences in Effects Between Men and Women
Brief Title: Prebiotic Effects of California Grapes on Gut Health and Cardiometabolic Health in Overweight Men and Women
Acronym: CALGRAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2172765; Proposal No 23-2586 (Other: California Table Grape Commission)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Arterial Stiffness; Blood Pressure; Dysbiosis; Inflammation; Permeability; Increased
Keywords: gut microbiome; nutrition; cardiometabolic health
MeSH Terms: conditions — Dysbiosis; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will limit intake of grapes and other polyphenol-rich foods while following their usual diet during the 1-week run-in period before the start of the intervention. They will be randomized to start with either grape or placebo powder for 3 weeks, consuming 48 grams of freeze-dried grape powder or placebo dissolved in water twice daily. Compliance will be assessed with three 24-hour dietary recalls using ASA24 and follow-up contact. After a 3-week washout period, participants will crossover to the other intervention. Study outcomes and anthropometry will be measured on the first and last days of each intervention arm, with the study lasting approximately 10-11 weeks for participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Freeze-dried grape powder or placebo powder packets labeled "A" and "1".
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape, Then Placebo (Experimental): Participants consume 48 grams of freeze-dried grape powder (dissolved into water) twice daily for 3 weeks. After a washout period of at least 3 weeks, participants then consume 48 grams of placebo powder matching grape powder (dissolved into water) twice daily for 3 weeks.
  Interventions: Dietary Supplement: Freeze-dried grape powder; Other: Placebo powder
- Placebo, Then Grape (Experimental): Participants consume 48 grams of placebo powder matching grape powder (dissolved into water) twice daily for 3 weeks. After a washout period of at least 3 weeks, participants then consume 48 grams of freeze-dried grape powder (dissolved into water) twice daily for 3 weeks.
  Interventions: Dietary Supplement: Freeze-dried grape powder; Other: Placebo powder

INTERVENTIONS:
Dietary Supplement: Freeze-dried grape powder — 48 grams powder
Other: Placebo powder — 48 grams powder

SUMMARY:
The goal of this clinical trial is to assess the impact of table grape consumption on gut microbiome, intestinal permeability, systemic inflammation, and vascular function in healthy overweight men and women aged 45-70 years. The main questions it aims to answer are:

* Does daily grape intake alter intestinal microbiome composition and intestinal permeability?
* Are changes in gut microbiota and intestinal permeability correlated with changes in cardiometabolic risk factors (inflammation, vascular function, lipid profiles)?
* Does response to grape intake on gut microbiota, intestinal permeability, cardiometabolic and inflammatory markers differ between men and women?
* Are metabolic pathways modified by grape consumption able to explain the link between gut health and cardiometabolic factors?

Researchers will compare freeze-dried grape powder to placebo powder to see if grape powder improves cardiometabolic risk factors.

Participants will

* Consume the powder dissolved in water twice daily for 3 weeks
* Follow their usual diet, modified to limit polyphenol-rich foods
* Visit the clinic at the beginning and end of the intervention for vascular measurements and blood sample collection
* Complete a 3-day 24-hour dietary recall and collect stool sample before each visit

DETAILED DESCRIPTION:
Participants will limit intake of grapes and other polyphenol-rich foods while following their usual diet during the 1-week run-in period before the start of the intervention. They will be randomized to start with either grape or placebo powder for 3 weeks, consuming 48 grams of freeze-dried grape powder or placebo dissolved in water twice daily. Compliance will be assessed with three 24-hour dietary recalls using ASA24 and follow-up contact. After a 3- to 4-week washout period, participants will crossover to the other intervention. Study outcomes and anthropometry will be measured on the first and last days of each intervention arm.

Aim 1: Biomarkers to assess the permeability of the gut, including zonulin, lipopolysaccharide (LPS), LPS-binding protein (LBP), soluble CD14, and diamine oxidase (DAO), will be analyzed from blood samples. Gut microbiome profiling will be analyzed from 16S rRNA gene sequencing of fecal samples collected by participants at the beginning and end of each intervention arm.

Aim 2: Vascular function will be assessed by measuring blood pressure and pulse wave velocity. After 15 minutes of rest, blood pressure will be measured three times, with the average of the latter two recorded. Pulse wave velocity from the carotid to femoral artery will measure arterial stiffness. Inflammatory cytokines will be assayed from blood samples to include Th17 cytokines. Lipid panel and comprehensive metabolic panels will also be analyzed.

Aim 3: Sex differences in response to grape consumption will be assessed, including gut microbiome, gut permeability, vascular function, inflammation, lipid profile, and metabolomic pathways. Gender and time interactions will be determined to assess differences in trajectory of changes.

Aim 4: LC-MS will be used for untargeted metabolomics and lipidomics. Pathway analysis will assess metabolic pathways affected by grape consumption and their links to gut permeability, systemic inflammation, and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women (cessation of menstruation for minimum two years)
* overweight and obese (BMI between 25-35 kg/m2)
* stable treatment for type 2 diabetes or metabolic syndrome
* ability to understand the intervention concept and written consent to participate
* willingness to accept randomization, undergo testing and intervention procedures, and deliver stool and blood samples

Exclusion Criteria:

* menopausal hormone replacement therapy started within less than 6 months
* antibiotics, prebiotics within last 3 months
* antidiabetic treatment involving insulin (for type 1 diabetes)
* vegetarian/vegan and not able to follow modified diet
* any serious medical condition including but not limited to coronary artery disease, uncontrolled hypertension, stroke, congestive heart failure, insulin-dependent diabetes, liver disease, active cancer and anemia
* psychiatric disease that interferes with the understanding and implementation of the intervention
* history of eating disorders such as bulimia nervosa, anorexia nervosa, severe binge eating disorder in the last 5 years
* history of substance abuse or alcohol abuse
* involvement in a weight loss intervention program (including anti-obesity medication) within last 3 months or have had bariatric surgery
* current smokers (within last 180 days)
* use of dietary supplements containing polyphenols in the past 1 month
* strenuous exercise greater than 10 hours per week

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Pulse Wave Velocity (PWV) from carotid to femoral artery after 5 minutes rest; PWV is an established index of aortic stiffness using a validated non-invasive device that allows online pulse wave recording and automatic PWV calculation
Blood pressure Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Average of latter 2 of 3 total measures (5 minutes apart) after 15 minutes of rest in a quiet room; SphygmoCor XCEL device will be used with participants in the seated position
Gut microbiome composition Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  16S rRNA sequencing of stool samples collected by participants from home in fecal collection tubes filled with DNA/RNA shield
Gut permeability markers Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  ELISA (zonulin, LPS, LBP, sCD14, DAO) to assay fasted blood samples collected when participants visit the clinic
Systemic inflammatory markers Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Luminex - Th17 inflammatory cytokines of fasted blood samples collected when participants visit the clinic
Lipid and metabolic profiles Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Lipid panel, comprehensive metabolic panel of fasted blood samples collected when participants visit the clinic

SECONDARY OUTCOMES:
Gut permeability marker Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  bacterial DNA presence in blood from fasted blood samples collected in tubes with DNA/RNA shield when participants visit the clinic
Metabolomics and Lipidomics Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Pathway Analysis using data available from analysis of blood samples collected when participants visit the clinic
Global gene expression Change from Baseline | Baseline (Visit 1), Week 3 (Visit 2), Week 9 (Visit 4)
  Microarrays of blood samples collected when participants visit the clinic

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Center, Davis, California, United States